CLINICAL TRIAL: NCT04442386
Title: Parental Burnout During the COVID-19 Pandemic: Risk Factors and Predictors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Collaborators: Modum Bad (Other)
Responsible Party: Principal Investigator, Omid V. Ebrahimi, Mr., University of Oslo
Other Study IDs: REK125510-15
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Parental Burnout
MeSH Terms: interventions — Prospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prospective study with two measurement points investigating the impact of viral mitigation protocols on parental burnout — Prospective study with two measurement points investigating the impact of viral mitigation protocols on parental burnout

SUMMARY:
The present study seeks to investigate the levels of parental burnout in the general parental population during the COVID-19 pandemic. Parental burnout is measured three months following (T2) the initiated viral mitigation protocols in Norway, a period where schools and kindergartens were closed, involving a period of home isolation for parents with their children. The burden of parents during this period is thought to have increased, as they were expected to conduct their own work virtually where possible, while at the same time acting as teachers for their children. The study aims to investigate the level of burnout among parents after months of viral mitigation strategies involved in the pandemic, in addition to predictors of parental burnout measured at (T1) are associated with parental burnout after three months (T2).

Hypothesis and research question:

Research Question 1: What is the level of parental burnout in the general parental population three months following initiated viral mitigation protocols (i.e., physical distancing) as compared to other similar pre-pandemic samples?

Hypothesis 1: Parental burnout will be higher in the present sample three months into the pandemic as compared to similar pre-pandemic samples in similar populations.

Hypothesis 2: Levels of parental stress, parental satisfaction, general self-efficacy, positive metacognitions, negative metacognitions, unhelpful coping strategies, marital quality and insomnia, all at T2 will significantly predict levels of parental burnout at T2.

Exploratory: Do the predictors parental stress, parental satisfaction, general self-efficacy, positive metacognitions, negative metacognitions, unhelpful coping strategies, all at baseline (T1), predict parental burnout at T2, beyond and above these same aforementioned predictors at T2 and pre-existing mental health condition, age, gender, and education?

Exploratory: Levels of parental burnout will be explored across subgroups in the sample.

DETAILED DESCRIPTION:
Hypothesis and research question:

Research Question 1: What is the level of parental burnout in the general parental population three months following initiated viral mitigation protocols (i.e., physical distancing) as compared to other similar pre-pandemic samples?

Hypothesis 1: Parental burnout will be higher in the present sample three months into the pandemic as compared to similar pre-pandemic samples in similar populations.

Hypothesis 2: Levels of parental stress, parental satisfaction, general self-efficacy, positive metacognitions, negative metacognitions, unhelpful coping strategies, marital quality and insomnia, all at T2 will significantly predict levels of parental burnout at T2.

Exploratory: Do the predictors parental stress, parental satisfaction, general self-efficacy, positive metacognitions, negative metacognitions, unhelpful coping strategies, all at baseline (T1), predict parental burnout at T2, beyond and above these same aforementioned predictors at T2 and pre-existing mental health condition, age, gender, and education?

Exploratory: Levels of parental burnout will be explored across subgroups in the sample.

Statistical analysis A hierarchical regression analysis will be conducted with Parental burnout (PBI) as the dependent variable. In the first step, stable characteristics (control variables) will be included: gender, education, and age. In the second step, parental stress, parental satisfaction, general self-efficacy, positive metacognitions, negative metacognitions, and unhelpful coping strategies, marital quality, and insomnia, all at T2 will be included.. In the final step, parental stress, parental satisfaction, general self-efficacy, positive metacognitions, negative metacognitions, and unhelpful coping strategies, all at T1 will be included.

Part correlations will be reported, presenting the effect size of the hypothesized predictors on parental burnout. A part (semi-partial) correlation gives the least biased and easiest interpretable estimate of the strength of a predictive relationship (Dudgeon, 2016). It is the correlation between the outcome and the aspects of the predictor unique from all the other predictors. As a type of correlation, its size can be evaluated according to Cohen's (1988) criteria: small >=0.10, medium >=0.30, large >=0.50.

Multicollinearity and other statistical assumptions will be checked. Multicollinearity will be assessed with common guidelines (VIF < 5 and Tolerance > 0.2; Hocking, 2003; O'Brian, 2007).

Descriptive statistics with frequency tables including N, means, SDs and other standard descriptive statistics will examine the research question concerning general levels of mental well-being. Subgroup differences will be examined.

All analyses and questions addressed in the forthcoming paper that are not pre-specified in this pre-registered protocol will be defined as exploratory.

Sensitivity analyses and random subsample replications of the main findings will be conducted following selection of a random sample of participants that ensure a proportionate ratio between the collected sample and the adult population of Norway.

Any questions addressed in the forthcoming paper which is not pre-specified in this protocol will be explicitly defined as exploratory.

Inference criteria Given the estimated large sample size which the investigators hope to collect in this study, the investigators pre-define their significance level: p < 0.01 to determine significance.

Sample size and power calculation:

The present study is part of a larger project with the first part aiming to investigate predictors of parental burnout through regression analyses, and the second part aiming to examine directional relations amongst specific symptoms and their centrality through complex systems approaches (i.e., network analysis). Consequently, power calculations are based on power required for network analyses. Following power analysis guidelines by Fried & Cramer (2017), it is recommended that the number of participants are three times larger than the number of estimated parameters. However, more conservative recommendations by Roscoe (1975) for multivariate research, recommends sample size that is ten times larger than the number of estimated parameters. Thus, following these two approaches respectively, between 900 to 3000 participants are required. Data will be collected for three weeks, and participants are based on a representative and random sample of Norwegian adults, randomly selected and provided equal opportunity to partake in the study, providing digital consent.

Missing data:

The TSD system (Services for Sensitive Data), a platform used in Norway to store person-sensitive data verifies participants officially through a kind of national ID number to give them full right to withdraw their data at any time, following the European GDPR (General Data Protection Regulation) laws. Accordingly, participants are allowed to withdraw their own data at any time. The survey includes mandatory fields of response. Participation is voluntarily, and withdrawal of provided data is possible at any moment. The investigators do not expect participants to withdraw their data and thus expect no missing data. However, if participants do withdraw their data, the investigators will conduct state-of-art missing data analyses and investigate whether data is missing at random.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are all parents
* Currently living in Norway and thus experiencing identical mitigation strategies
* That provide digital consent to partake in the study

Exclusion Criteria:

* Adults not residing in Norway during the measurement period
* Non-parents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both Biological Sex and self-representation of gender are measured
Study Population: All parents above 18 years residing in Norway and thus experiencing identical mitigation protocols are invited to participate the study, reaching randomly online with an equal opportunity of participating.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-06-22 (Estimated); Primary Completion 2020-07-13 (Estimated); Study Completion 2020-07-13 (Estimated)

PRIMARY OUTCOMES:
The Parental Burnout Inventory (PBI) | Data is set to be collected starting from 22nd of June until enough data has been collected. The data collection period will last no longer than three weeks
  The Parental Burnout Inventory (PBI) (Roskam et al., 2017) consists of 22 items related to three divisions of parental burnout: Personal Accomplishment, Emotional Exhaustion and Emotional Distancing. The inventory is rated on a seven-point Likert-scale ranging from never (0) to every day (6). Higher scores indicate greater parental burnout severity, and scores above 88 are considered as the cut-off for parental burnout (Roskam et al., 2017).

CONTACTS AND LOCATIONS:
Overall Officials: Nora Paulsen Skjerdingstad, Cand.psychol. stud, Principal Investigator — University of Oslo; Miriam Sinkerud Johnson, PhD, Principal Investigator — Oslo Metropolitan University; Sverre Urnes Johnson, PhD, Principal Investigator — University of Oslo; Asle Hoffart, PhD, Principal Investigator — Modum Bad; Omid V. Ebrahimi, Double PhD Candidate, Principal Investigator — University of Oslo

REFERENCES:
- [Background] Roskam I, Raes ME, Mikolajczak M. Corrigendum: Exhausted Parents: Development and Preliminary Validation of the Parental Burnout Inventory. Front Psychol. 2018 Jan 30;9:73. doi: 10.3389/fpsyg.2018.00073. eCollection 2018. PMID 29403419